CLINICAL TRIAL: NCT00031460
Title: A Placebo-Controlled Phase III Evaluation of Suppressive Therapy With Oral Acyclovir Suspension Following Neonatal Herpes Simplex Virus Infections Involving the Central Nervous System
Brief Title: Acyclovir for Herpes Infections Involving the Central Nervous System in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 97-007; CASG 103; N01AI30025C; N01AI30025 (NIH); NCT00000934 (obsolete NCT alias)
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2009-10

CONDITIONS: Herpes Simplex
Keywords: acyclovir, central nervous system, Herpes Simplex Virus
MeSH Terms: conditions — Herpes Simplex | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Acyclovir (Experimental)
  Interventions: Drug: Acyclovir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir — Oral banana flavored acyclovir suspension: 300 mg/m^2/dose three times a day (TID), to be given at least 6 to 8 hours apart for 6 months. Dosage adjustments will be made monthly to compensate for increases in body surface area.
  Arms: Acyclovir
Drug: Placebo — Oral banana flavored placebo suspension: to be given at least 6 to 8 hours apart for 6 months. Dosage adjustments will be made monthly to compensate for increases in body surface area.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether long term treatment with acyclovir given orally (by mouth) improves the outcome for infants with herpes simplex virus infection of the brain or spinal cord (known as the central nervous system [CNS]). Infants with herpes viral infection of the CNS that has or has not spread to other parts of the body will be enrolled in this study. All participants will receive treatment in a hospital for 21 days with acyclovir, given intravenously (by a needle inserted into a vein). Participants will then be divided into two groups: those with CNS disease that has or has not spread to the skin, and those whose viral infection has spread and involves the CNS. Both groups will be randomly assigned to receive either oral acyclovir or placebo (inactive substance) for 6 months. Infants in the US and Canada will participate for 5 years. A physical exam, hearing exam, eye exam, and an evaluation of the nervous system will be performed throughout the study.

DETAILED DESCRIPTION:
Neonatal herpes simplex virus (HSV) disease complicates approximately 1 in every 3,000 deliveries in the United States, resulting in an estimated 1, 500 cases annually in this country. HSV-1 and HSV-2 infections in the neonate can manifest as: disseminated disease; central nervous system (CNS) disease; or disease limited to the skin, eyes, and mouth (SEM disease). This study will evaluate the efficacy of long term suppressive therapy with oral acyclovir in infants with CNS disease, with or without evidence of dissemination to other organs (including the skin). It will determine if suppressive oral acyclovir therapy improves neurologic outcome in infants following HSV disease with CNS involvement and address the significance of a positive cerebral spinal fluid (CSF) polymerase chain reaction (PCR) result when all other CSF parameters either remain normal or show improvement. Comparisons will be made between groups with respect to post-randomization time to first positive CSF PCR result during the initial 12 months of life, and results will be correlated with clinical neurological assessments. It will determine if continuous administration of oral acyclovir suspension suppresses recurrent skin lesions in infants following HSV disease with CNS involvement, and it will confirm the safety of long-term administration of oral acyclovir therapy in a cohort of infants with HSV disease with CNS involvement. Finally, the effects of suppressive acyclovir therapy on issues of pharmacoeconomics and family infrastructure will be assessed and quantitated. Infants with CNS disease (with or without evidence of viral dissemination to other organs, such as the skin, liver, and lungs) will qualify for this study. Following a 21 day course of treatment with intravenous (IV) acyclovir, infants with CNS disease, with or without cutaneous involvement, will be randomized to either continuous oral acyclovir or placebo (CNS Sub-Study). Similarly, infants with disseminated disease with CNS involvement will be randomized to either continuous oral acyclovir or placebo (Disseminated with CNS Involvement Sub-Study). The subset of infants with CNS disease (with or without dissemination) who do not clear their acute infection in 21 days of IV acyclovir therapy will be eligible for enrollment in a Pilot Sub-Study. This group is expected to be of insufficient number to be able to obtain statistical significance for establishing efficacy. Per protocol amendment dated 19-Nov-1998, 66 subjects will be recruited into each sub-study. Subjects will begin oral drug therapy 8 hours after the final IV acyclovir dose and oral drug therapy will be administered for 6 months. Whole blood (1.0 cubic centimeter) will be obtained at study enrollment and at completion of IV antiviral therapy for HSV PCR analysis, per protocol amendment dated 4-May-1998. This amendment replaces the obtaining of serum for HSV PCR analysis. In the event that whole blood is not available, serum will be provided instead. All children will be followed at 6, 12, 24, 36, 48, and 60 months of age. Physical examination, hearing assessment, and retinal examination will be performed at each follow-up visit. Standardized neurological evaluations will be performed at 12, 24, 36, 48, and 60 months. The primary study endpoint will evaluate neurological impairment at 12 months of life. The secondary endpoints will evaluate post-randomization detection of HSV DNA in CSF by PCR at any time during the initial 12 months of life and 2 or fewer episodes post-randomization of cutaneous recurrence of HSV disease during the initial 12 months of life.

ELIGIBILITY:
Inclusion Criteria:

* Viral Culture:

  1. If cutaneous lesions are present, then isolation of Herpes Simplex Virus (HSV)-1 or HSV-2 by viral culture from any site (skin, oropharynx, cerebral spinal fluid [CSF], urine, etc.) will be required for study entry.
  2. If cutaneous lesions are not present, then viral isolation by culture is adequate for study entry but is not required. In the case of no cutaneous lesions and negative viral cultures, however, the CSF polymerase chain reaction (PCR) must be positive.
  3. Additional sites from which HSV culture will be attempted include conjunctivae, oropharynx, blood buffy coat, urine, and CSF.
* Evidence for central nervous system (CNS) HSV disease during the acute illness, including one or more of the following:

  1. Abnormal CSF indices for term infants: greater than 22 white blood cells (WBCs)/mm^3 and protein greater than 115mg/dl.
  2. Abnormal CSF indices for preterm infants: greater than 25 WBCs/mm^3 and protein greater than 220 mg/dl.
  3. Abnormal neuroimaging study (computed tomography [CT] with contrast, magnetic resonance imaging [MRI] with gadolinium, or head ultrasound) [NOTE: CT with contrast is the preferred imaging study].
  4. Abnormal electroencephalography (EEG), if performed (NOTE: EEG is suggested for the evaluation of infants with HSV disease but is not required for this study].
  5. Positive CSF PCR for HSV deoxyribonucleic acid (DNA) [NOTE: If no cutaneous lesions are present and all viral cultures are negative, the CSF PCR must be positive. If lesions are present and are culture-positive, abnormal CNS neurodiagnostic studies or abnormal CSF indices are sufficient for study entry].
* Negative CSF PCR result within 48 hours prior to completion of intravenous acyclovir therapy.
* Less than or equal to 28 days of age at the time of initial presentation with CNS disease.
* Birth weight greater than or equal to 800 grams.

Exclusion Criteria:

* Infants with either a grade 3 or grade 4 intraventricular hemorrhage (IHV) prior to study enrollment.
* Breast feeding infants whose mothers are taking acyclovir, valacyclovir, or famciclovir for greater than 120 hours (greater than 5 days). If at any point following enrollment the mother takes these antiviral drugs for greater than 120 hours (greater than 5 days), she will be asked to refrain from breast feeding while taking the drug.
* Infants known to be born to women who are human immunodeficiency virus (HIV) positive (but HIV testing is not required for study entry). These infants are at known risk of acquiring HIV, which would alter their immune response to other infections, including herpes simplex virus (HSV) infection. Additionally, they may be receiving antiretroviral and/or antiviral drugs during the time in which the study of suppressive oral acyclovir is being conducted. As such, they will be excluded if the mother's positive HIV status is known at the time of evaluation for study inclusion. If at any point following enrollment it is learned that an infant is HIV positive, however, he/she will be continued on the study protocol.
* Infants with HSV infection limited to the skin, eyes, or mouth (SEM). Patients with SEM HSV infection will be considered for enrollment and randomization in the ongoing Collaborative Antiviral Study Group (CASG) evaluation of oral suppressive acyclovir therapy following neonatal HSV infections limited to the SEM.
* Infants with creatinine greater than 1.5 mg/dl at time of study enrollment.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 1997-12; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Department of Infectious Diseases, Little Rock, Arkansas
  - Children's Hospital Los Angeles - Pediatrics Infectious Diseases, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - University of Florida - College of Medicine - Jacksonville, Jacksonville, Florida
  - The University of Chicago - Comer Children's Hospital - Infectious Diseases, Chicago, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University - Tulane Medical Center - Department of Pediatrics, New Orleans, Louisiana
  - Maine Medical Center - Department of Pediatric Specialty Care - Infectious Disease, Portland, Maine
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital of Michigan - Pediatric Infectious Diseases, Detroit, Michigan
  - University of Mississippi, Jackson, Mississippi
  - St. Louis Children's Hospital - Infectious Disease, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - UNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center - Pediatric Infectious Disease, Cleveland, Ohio
  - Nationwide Children's Hospital - Infectious Diseases, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Infectious Disease Services, Fort Worth, Texas
  - University of Texas Health Science Center San Antonio - Pediatrics - Immunology & Infectious Disease, San Antonio, Texas
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington
- University of Alberta - Aberhart Centre - Pediatrics, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Kimberlin DW, Whitley RJ, Wan W, Powell DA, Storch G, Ahmed A, Palmer A, Sanchez PJ, Jacobs RF, Bradley JS, Robinson JL, Shelton M, Dennehy PH, Leach C, Rathore M, Abughali N, Wright P, Frenkel LM, Brady RC, Van Dyke R, Weiner LB, Guzman-Cottrill J, McCarthy CA, Griffin J, Jester P, Parker M, Lakeman FD, Kuo H, Lee CH, Cloud GA; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Oral acyclovir suppression and neurodevelopment after neonatal herpes. N Engl J Med. 2011 Oct 6;365(14):1284-92. doi: 10.1056/NEJMoa1003509. PMID 21991950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neonates diagnosed with HSV-1 or HSV-2 <= 28 days of age with evidence of CNS HSV disease (with or without evidence of viral dissemination to other organs, such as the skin, liver, and lungs) then treated with intravenous acyclovir therapy. Subject has negative CSF PCR results within 48 hours prior to completion of intravenous acyclovir therapy.
Pre-assignment Details: Subjects enrolled while on 2 - 3 weeks of IV acyclovir therapy who have positive cerebrospinal Fluid (CSF) herpes simplex virus (HSV) PCR results within 48 hours prior to IV therapy completion, are not randomized.
Groups:
- Acyclovir: Oral suspension 300 mg/m^2/dose TID for 6 months.
- Placebo: Identical volume as acyclovir.
Period: Overall Study
Arm/Group | Acyclovir | Placebo
Started | 24 | 22
Completed | 15 | 8
Not Completed | 9 | 14
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Non-Compliant | 1 | 1
Not completed — Death | 0 | 1
Not completed — Reactivation of Disease | 5 | 9
Not completed — Disruption of blinded drug supply | 2 | 0
Not completed — Confirmed unevaluable | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyclovir | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Customized [Median (Full Range); unit: days] | 11 (1.71) [1 to 42] | 15.5 (1.42) [5 to 29] | 13 (1.13) [1 to 42]
Age, Customized [Number; unit: participants]
  <=28 days | 24 | 22 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43
  Canada | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Participants With Neurologic Impairment at 12 Months as Measured by a Bayley's Neuro-developmental Assessment (Motor Scores).
Description: Motor scores of all participants completing 6 months of blinded therapy as measured by the Bayleys neuro-developmental assessment at 12 months. Scores are classified as the following: greater than or equal to 115 suggests accelerated performance; 85 - 114 suggests development within normal limits; 70 - 84 suggests mildly delayed development; and less than or equal to 69 suggests significant delayed development.
Time Frame: At 12 months of life.
Measure: Number; unit: participants
Arm/Group | Acyclovir | Placebo
Number analyzed (Participants) | 15 | 8
participants
  Units: participants | 10 | 5
  Number of participants with score > or = 115 | 0 | 1
  Number of participants with score 85 - 114 | 6 | 2
  Number of participants with score 70 - 84 | 0 | 0
  Number of participants with score< or = 69 | 4 | 2

2. Secondary Outcome: Number of Participants With Two or Fewer Episodes of Cutaneous Recurrence of Herpes Simplex Virus (HSV) Disease Post-randomization During the Initial 12 Months of Life.
Description: Number of participants experiencing 2 or fewer HSV recurrences during the first 12 months of life as measured by assessments and reports at study visits.
Time Frame: post randomization - 12 months
Measure: Number; unit: participants
Arm/Group | Acyclovir | Placebo
Number analyzed (Participants) | 15 | 8
participants
  Number of participants reporting recurrences | 6 | 3
  Participants with < or = 2 recurrences | 3 | 1
  Participants with > 2 recurrences | 3 | 2

3. Secondary Outcome: Detection of Herpes Simplex Virus (HSV) DNA in the Cerebrospinal Fluid (CSF) by PCR at Anytime During the Initial 12 Months of Life.
Description: Number of participants assessed to have a positive herpes simplex virus (HSV) DNA by polymerase chain reaction (PCR) in the cerebrospinal fluid (CSF) at any time during their initial 12 months of life after treatment. The PCR is a technique to help visualize copies of a piece of DNA.
Time Frame: post randomization - 12 months
Measure: Number; unit: participants
Arm/Group | Acyclovir | Placebo
Number analyzed (Participants) | 15 | 8
participants
  Number of participants reporting = or >1 + CSF PCR | 12 | 6
  Number of participants reporting 0 - CSF PCR | 3 | 2

4. Primary Outcome: Participants With Neurologic Impairment at 12 Months as Measured by Bayley's Neuro-developmental Assessment.(Mental Scores)
Description: Mental scores of all subjects completing 6 months of blinded therapy as measured by the Bayleys neuro-developmental assessment at 12 months. Scores are classified as the following: greater than or equal to 115 suggests accelerated performance; 85 - 114 suggests development within normal limits; 70 - 84 suggests mildly delayed development; and less than or equal to 69 suggests significant delayed development.
Time Frame: At 12 months of life.
Measure: Number; unit: participants
Arm/Group | Acyclovir | Placebo
Number analyzed (Participants) | 15 | 8
participants
  Number of participants reporting scores | 10 | 6
  Participants with score > or = 115 | 0 | 1
  Participants with score 85 - 114 | 7 | 1
  Participants with score 70 - 84 | 0 | 0
  Participants with score < or = 69 | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were followed throughout the 5 years of the study subject participation, or until subject terminated from the study. Subjects not completing 6 months of study drug were followed as intent to treat.
Description: Twenty-two participants were enrolled into the placebo arm; however, only 21 received study drug.
Arm/Group | Acyclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 17/24 | 15/21
Other Adverse Events (participants affected / at risk) | 18/24 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir (N=24) | Placebo (N=21)
Decreased neutrophils (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Feeding dysfunction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 2 (2) | 0 (0)
Herpes simplex virus (Infections and infestations) | 4 (5) | 8 (13)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 3 (3)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Infantile spasms (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir (N=24) | Placebo (N=21)
Neutropenia (Blood and lymphatic system disorders) | 11 (17) | 4 (4)
Herpes simplex virus (Infections and infestations) | 6 (21) | 8 (26)
Otitis media (Infections and infestations) | 7 (10) | 8 (12)
Upper respiratory infection (Infections and infestations) | 7 (12) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No